CLINICAL TRIAL: NCT05640076
Title: Effects of a 24/7 Palliative Care Service Integration in a Metropolitan Area on Non-oncologic Patients
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: FEDERATION
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Palliative Medicine; Hospice and Palliative Care Nursing; Palliative Care
Keywords: Medicine, Palliative; Palliative Care; Hospice and Palliative Care Nursing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 2018-19 - Oncologic patients under home palliative care: Oncologic patients took over from the Metropolitan Palliative Care Service and receiving home palliative care within their last 90 days of life between 1/1/2018 and 31/12/2019
  Interventions: Other: 24/7 Telephonic Palliative Care Service availability
- 2018-19 - Non-oncologic patients under home palliative care: Non-oncologic patients took over from the Metropolitan Palliative Care Service and receiving home palliative care within their last 90 days of life between 1/1/2018 and 31/12/2019
- 2021-2022 - Oncologic patients under home palliative care: Oncologic patients took over from the Metropolitan Palliative Care Service and receiving home palliative care within their last 90 days of life between 1/1/2021 and 31/12/2022
  Interventions: Other: 24/7 Telephonic Palliative Care Service availability
- 2021-2022 - Non-Oncologic patients under home palliative care: Non-oncologic patients took over from the Metropolitan Palliative Care Service and receiving home palliative care within their last 90 days of life between 1/1/2021 and 31/12/2022
  Interventions: Other: 24/7 Telephonic Palliative Care Service availability

INTERVENTIONS:
Other: 24/7 Telephonic Palliative Care Service availability — Metropolitan Palliative Care Service-implemented 24/7 telephonic availability service for the patients, their relatives, the EMS and Primary Care physicians taking care of them.
  After consultation, if the information and medical suggestions are not sufficient, an urgent ambulatory or home visit could be planned.
  Groups: 2018-19 - Oncologic patients under home palliative care; 2021-2022 - Non-Oncologic patients under home palliative care; 2021-2022 - Oncologic patients under home palliative care

SUMMARY:
This retrospective observational pre-post study aims to test the effects of introducing a remote telephonic consultation availability from the Palliative Care Service for a cohort of non-oncologic patients followed by the same service, their relatives, and the Emergency Medical Services (EMS) and family care physicians taking care of them.

The main question[s] it aims to answer are:

* Does the introduction of a remote telephonic consultation availability affect the rate of ED access of non-oncologic Palliative-care followed patients during their last 90 days of life?
* Does the introduction of a remote telephonic consultation availability have an effect on the rate of EMS requests for these patients during their last 90 days of life?
* Which are the main topics of the calls to the Palliative Care Service?

Due to the emergence of COVID-19 pandemic during the study period, a parallel cohort of oncologic patients under 24/7 palliative care by the same service during both the observation periods will be used as reference.

Participants will be followed up from the date of taking-over request to the Palliative Care Service to their death or the end of the period of observation if followup began during their last 90 days of life.

Otherwise, for those being already under home palliative care at the 90th day before their death, follow up will begin at that day.

Researchers will compare two time periods to see if the introduction of a remote telephonic consultation availability has an effect on the supra-mentioned aims.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed by the Metropolitan Palliative Care Service of Bologna
* Residency in Bologna Metropolitan city

Exclusion Criteria:

* Incomplete data
* Residency outside Bologna Metropolitan City

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in the study is composed of the whole population of patients followed by the palliative care metropolitan service of Bologna respecting the Eligibility criteria shown
Sampling Method: Probability Sample
Enrollment: 2831 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Emergency Department Admission rate of patients followed by the Palliative Care Service | 48 months

SECONDARY OUTCOMES:
EMS calls rate from patients followed by the Palliative Care Service | 48 months
Main topics of the calls received from the Palliative Care Service after the full implementation of a 24/7 service | 24 months
  Classification of the topics of the calls into 5 main classes: "Clinical questions", "Caregiver Support", "Definition of care pathway", "Palliative sedation", "Other communications".
  The relative frequency of each main topic will be reported

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Unità Sanitaria Locale, Bologna
  - IRCCS - Policlinico Universitario S.Orsola - Malpighi, Bologna

IPD SHARING:
Plan to Share IPD: No
IPD will be shared if requested under appropriate motivation

REFERENCES:
- [Background] Burge F, Lawson B, Johnston G. Family physician continuity of care and emergency department use in end-of-life cancer care. Med Care. 2003 Aug;41(8):992-1001. doi: 10.1097/00005650-200308000-00012. PMID 12886178
- [Background] Barbera L, Paszat L, Chartier C. Indicators of poor quality end-of-life cancer care in Ontario. J Palliat Care. 2006 Spring;22(1):12-7. PMID 16689410
- [Background] Gamblin V, Prod'homme C, Lecoeuvre A, Bimbai A-, Luu J, Hazard PA, Da Silva A, Villet S, Le Deley MC, Penel N. Home hospitalization for palliative cancer care: factors associated with unplanned hospital admissions and death in hospital. BMC Palliat Care. 2021 Jan 26;20(1):24. doi: 10.1186/s12904-021-00720-7. PMID 33499835
- [Background] Thomsen JL, Parner ET. Methods for analysing recurrent events in health care data. Examples from admissions in Ebeltoft Health Promotion Project. Fam Pract. 2006 Aug;23(4):407-13. doi: 10.1093/fampra/cml012. Epub 2006 Apr 4. PMID 16595540
- [Derived] Valenti D, Gamberini L, Allegri D, Tartaglione M, Moggia F, Del Giudice D, Baroni R, Di Mirto CVF, Tamanti J, Rosa S, Paoletti S, Bruno L, Peterle C, Cuomo AMR, Bertini A, Giostra F, Mengoli F; Collaborators. Effects of 24/7 palliative care consultation availability on the use of emergency department and emergency medical services resources from non-oncological patients: a before-and-after observational cohort study. BMJ Support Palliat Care. 2024 Dec 19;14(e3):e2788-e2797. doi: 10.1136/spcare-2023-004412. PMID 37973206